CLINICAL TRIAL: NCT00730678
Title: Pharmacogenetic Determinants Of Treatment Response In Children
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: PGEN5; R37CA036401 (NIH); P50GM115279 (NIH); R01CA036401 (NIH); R01GM118578 (NIH); R35GM141947 (NIH); R01CA264837 (NIH); NCI-2021-09904 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: All Malignancies; Children Being Treated for Catastrophic Illness
Keywords: Metabolism; Pharmacogenetic testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA or RNA for genetic testing will typically be obtained simultaneously with blood that is drawn for clinical reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants enrolled on this study will have blood drawn for genetic testing.

SUMMARY:
To investigate whether genetic polymorphisms in genes encoding proteins involved in the metabolism or effects of drugs or environmental agents influence the disposition or effects of these xenobiotic substrates. To investigate the nature of heritability and the genetic basis of pharmacogenetic traits by studying family members of individuals with specific genotypes.

DETAILED DESCRIPTION:
Pharmacogenetics is that discipline devoted to elucidating the genetic determinants of drug response. Particularly in the area of drug metabolism, many genes exhibit genetic polymorphism; that is, a stable percentage of the population (which generally differs by ethnic group) is deficient in the functional expression of the enzyme involved, and the deficiency is typically inherited as an autosomal recessive trait. With currently known polymorphisms in drug metabolism, the percentage of homozygous deficient individuals ranges from 0.3% to as many as 90% of the population, depending on the enzyme and the ethnic group.

Our prior studies have revealed multigenic pharmacogenetic models that are significantly predictive of various drug response phenotypes (e.g., drug resistance, drug clearance, drug toxicity, disease response) in children with ALL. The large number of candidate loci and the relatively small number of patients illustrate the fact that larger sample sizes are required to definitively establish these polygenic models. The fact that there were significant race/genotype interactions, such that predictions differed in whites vs blacks, highlights the need for adequate numbers of patients within racial and ethnic groups to allow differential analysis of genotypic predictors after adjusting for confounding demographic factors in pharmacogenetic studies via stratified design and analyses.

ELIGIBILITY:
Inclusion Criteria:

* Any patients under evaluation/treatment at St. Jude Children's Research Hospital (SJCRH)
* Parents or family members of St. Jude patients
* Non patient volunteers
* All study subjects must provide informed consent for participation
* Assent/Consent of the patient (parent) must be provided prior to attempts made by investigators to enroll a family member of a SJCRH patient

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated at St. Jude Children's Research Hospital are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8800 (Estimated)
Dates: Start 1998-08-17 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
To investigate whether genetic polymorphisms in genes encoding proteins involved in the metabolism or effects of drugs or environmental agents influence the disposition or effects of these xenobiotic substrates. | 28 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun J Yang, Ph. D., Principal Investigator — St. Jude Children's Research Hospital; Kristine Crews, PharmD, MSCI, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols